CLINICAL TRIAL: NCT02767427
Title: The Value of Home Chlorhexidine Pre-Surgical Wash Before Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Orthopaedic Scientific Research Foundation Inc (Unknown)
Responsible Party: Principal Investigator, Kiehyun Riew, Professor of Orthopedic Surgery at the Columbia University Medical Center, Columbia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AAAP8304
Record Dates: First submitted 2016-04-23; First posted 2016-05-10 (Estimated); Results first posted 2019-07-16 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Infection; Spinal Injuries
Keywords: Infection Control; Preoperative Care; Chlorhexidine; Pre-Surgical Wash; Spine Surgery; Surgical site infections; Cutaneous bacterial load on skin
MeSH Terms: conditions — Infections; Spinal Injuries; Surgical Wound Infection

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- At-Home Chlorhexidine (Active Comparator): Those randomized into the chlorhexidine group will be asked to shower the night before surgery, and to use a standardized pre-packaged Chlorhexidine Wipes (chlorhexidine gluconate wipes) on their surgical site after thoroughly drying those areas. They will be asked to use a second wipe in each area the morning of surgery. Those who forget to use the wipe in the morning were allowed to use the wipe in the pre-operative area and included if this occurs more than one hour before skin prep.
  Interventions: Device: Chlorhexidine Wipes
- No At-Home Chlorhexidine (Experimental): Participants in this group will not use chlorhexidine wipes (no intervention), as is standard of care, prior to their surgical site being cleansed by the surgical team pre-operatively.
  Interventions: Other: No intervention

INTERVENTIONS:
Device: Chlorhexidine Wipes — (Standard of Care) Chlorhexidine wipes are a commonly used pre-operative skin cleansing measure, designed to reduce bacterial load on the skin of the surgical site.
  Other Names: 4% Chlorhexidine Wipes; Chlorhexidine Gluconate; Skin Prep Cloths; Sage Skin Prep Cloths
  Arms: At-Home Chlorhexidine
Other: No intervention — Chlorhexidine wipes will not be used though it is a commonly used pre-operative skin cleansing measure.
  Arms: No At-Home Chlorhexidine

SUMMARY:
The study team hypothesizes that at-home cleansing of the surgical site with chlorhexidine wipes provide no added benefit to decreasing microbial activity or preventing surgical site infections.

Patients will be randomized to the chlorhexidine or no additional intervention groups. Patients will be randomized to use 4% chlorhexidine cloths, while the other half receive no additional intervention. Those randomized into the chlorhexidine gluconate (CHG) home-application group will be asked to shower the night before surgery, and to use a standardized pre-packaged CHG wipe (that the patients would receive at their pre-surgical consultation) on their surgical site after thoroughly drying those areas. The patients will be asked to use a second wipe in each area the morning of surgery. The surgical sites will be analyzed in two groups: anterior cervical and posterior spine. Each of these two groups will be randomized separately. All patients will undergo a standardized preoperative cleansing regimen. Once positioned, they will be cleansed with an alcohol solution. Then, the surgical site (either the anterior portion of the neck or the posterior area of the spine) will be scrubbed with chlorhexidine soaked brushes and then painted with chlorhexidine solution. Perioperative antibiotics will be given per attending surgeon preference. Cutaneous samples will be taken from the surgical site of each patient at each time point.

DETAILED DESCRIPTION:
To the investigator's knowledge no prior study has evaluated the effects of cleaning the skin at home before surgery in patients undergoing spine surgery. This study will investigate whether patients who use a chlorhexidine cleansing wipe have decreased amounts of bacteria on their skin when they arrive for scheduled spine surgery. Spine surgeons strive to decrease infections in their patients, so it is important to see if this intervention helps to do this.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Scheduled for elective spine surgery at Columbia University Medical Center

Exclusion Criteria:

* Unable to apply at-home chlorhexidine wipe by themselves
* Deemed "high risk" preoperatively by the treating surgeon
* Diagnosed with spine trauma
* Undergoing deformity correction surgery
* Unable to consent to the terms of the surgery
* Known infection at time of the index procedure
* Hospitalized within 1 week pre-operatively
* Allergic to chlorhexidine
* Immunocompromised
* End stage renal disease on dialysis
* Local or systemic skin disease (such as psoriasis, eczema, etc.)
* Open skin wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kiehyun D Riew, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | At-Home Chlorhexidine | No At-Home Chlorhexidine
Started | 21 | 19
Completed | 21 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- At-Home Chlorhexidine: Those randomized into the chlorhexidine group will be asked to shower the night before surgery, and to use a standardized pre-packaged Chlorhexidine Wipes (chlorhexidine gluconate (CHG) wipes) on their surgical site after thoroughly drying those areas. They will be asked to use a second wipe in each area the morning of surgery. Those who forget to use the wipe in the morning were allowed to use the wipe in the pre-operative area and included if this occurs more than one hour before skin prep.
  Chlorhexidine Wipes: (Standard of Care) Chlorhexidine wipes are a commonly used pre-operative skin cleansing measure, designed to reduce bacterial load on the skin of the surgical site.
- Total: Total of all reporting groups
Arm/Group | At-Home Chlorhexidine | No At-Home Chlorhexidine | Total
Number analyzed (Participants) | 21 | 19 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 12 | 30
  >=65 years | 3 | 7 | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.05 (9.12) | 59.79 (13.10) | 57.87 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 14 | 13 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 19 | 14 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 19 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Cutaneous Bacterial Load After Surgery
Description: All specimens were taken by a sterile BD E-Swab. All samples will be sent immediately after acquisition to the microbiology lab for analysis within four hours.
Time Frame: Pre-Surgery and Post Surgery, up to 4 hours
Measure: Count of Participants; unit: Participants
Arm/Group | At-Home Chlorhexidine | No At-Home Chlorhexidine
Number analyzed (Participants) | 21 | 19
Participants
  Presurgery Bacterial Colony Count: Subjects with bacterial colonies | 0 | 18
  Presurgery Bacterial Colony Count: Subjects without bacterial colonies | 21 | 1
  Postsurgical Bacterial Colony Count: Subjects with bacterial colonies | 0 | 0
  Postsurgical Bacterial Colony Count: Subjects without bacterial colonies | 21 | 19
Statistical Analysis 1: Comparison: At-Home Chlorhexidine vs No At-Home Chlorhexidine; Test type: Equivalence — An equivalence test on data from a parallel-group design with sample sizes of 18 in the reference group and 18 in the treatment group achieves 80% power. The significance was set at 5%. The standard deviation was 1.00, and the equivalence limits were set at -1.00 and 1.00; p < 0.05, t-test, 1 sided; Two one-sided t-tests were conducted with 18 in each group

ADVERSE EVENTS:
Time Frame: The forty enrolled patients were all consented and followed for data collection over the span of 15 months. Each patient was followed for up to 6 weeks after surgery to ensure that there were no postoperative infections.
Arm/Group | At-Home Chlorhexidine | No At-Home Chlorhexidine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/19
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/19
Other Adverse Events (participants affected / at risk) | 0/21 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/27/NCT02767427/Prot_SAP_000.pdf